CLINICAL TRIAL: NCT02934581
Title: Prevalence Rate, and Clinical Characteristics of Obesity Hypoventilation Syndrome Via Screening Patients Admitted to Medical Intensive Care Units
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201409020RINC
Record Dates: First submitted 2016-09-20; First posted 2016-10-17 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2016-10

CONDITIONS: Obesity Hypoventilation Syndrome
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective observation study to screen adult obese (BMI ≥30 kg/m2) patients who were newly admitted to the medical intensive care units and turned out to be diagnosed as Obesity hypoventilation syndrome(OHS). The investigators purpose is to look into the prevalence, predictive factors, and outcomes of OHS in these critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m2
* Suspected chronic hypercapnia as following Paco2 ≥ 45 mmHg, HCO3- ≥ 27mEq/L or base excess, BE ≥ 2 mEq/L

Exclusion Criteria:

* Malignancy with lung involvement
* Autoimmune disease with lung involvement
* Moderate to severe obstructive respiratory pattern via spirometry
* Uncontrolled endocrine disease
* Pregnancy
* Pneumonia confirmed by image
* Out-of-hospital cardiac arrest
* Lung edema
* Foreigner of Taiwan

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult obese (BMI ≥30 kg/m2) patients who were newly admitted to the medical intensive care units and turned out to be diagnosed as obesity hypoventilation syndrome
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-10-29 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of obesity hypoventilation syndrome in Asian critically ill patients | 2-year
  Detecting obesity hypoventilation syndrome via screening obesity(BMI>=30kg/m^2) in critical care units in Asian.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided